CLINICAL TRIAL: NCT05629169
Title: Video Review of the Frequency and Assessment of Head Impacts During the FIFA World Cup 2022TM
Status: Completed | Type: Observational
Sponsor: Federation Internationale de Football Association (Other)
Collaborators: Major League Soccer (Unknown)
Responsible Party: Sponsor
Other Study IDs: 004
Record Dates: First submitted 2022-11-17; First posted 2022-11-29 (Actual); Last update posted 2025-02-11 (Actual); Status verified 2024-03

CONDITIONS: Head Injury; Concussion; Brain Injuries; Traumatic Brain Injury
MeSH Terms: conditions — Craniocerebral Trauma; Brain Concussion; Brain Injuries; Brain Injuries, Traumatic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: No intervention applied - observational study only — Observational study only. All head impacts will be assessed using video footage.

SUMMARY:
This is an exploratory observational study.

Broadcasted video footage is used to review all head impacts during all 64 matches in the football tournament.

All head impacts are registered, and simple descriptive statistics are used to create overviews of the head impact characteristics, including video signs of potential concussion, observed contact, location of the head impact, presence and timing of medical assessment, whether there was foul play and sanction, and if the player was substituted.

DETAILED DESCRIPTION:
This study will be performed at the FIFA World Cup 2022, a football tournament including 32 national men's senior football teams. The tournament includes 64 matches played in Qatar between November 20th and December 18th, 2022.

Recording of head impacts The investigators will use injury spotters and subsequent video footage review to study head impacts. All matches will be attended by one of eight FIFA injury spotters, who will register all head impacts on a standardized scoring form. All FIFA injury spotters are qualified medical doctors with experience in football medicine and are also FIFA Medical Coordinators in other matches at the same tournament. The injury spotters are positioned on the tribune above the midline of the pitch with visibility of the entire pitch. If the injury spotter observes a head impact, they can review video footage on a large computer screen immediately to identify possible mechanism of injury and the presence of video signs indicating a possible concussion. The injury spotter can select one or more angles for review at the same time (up to four close views and four wide views) and rewind and forward at different speeds, including frame-to-frame views.

A modification of a previous definition of a head impact was clarified to: "a direct head impact, or impact with indirect forces to the head, where a player is unable to immediately resume play following impact or subsequently shows potential concussion-related symptoms."

Video signs The investigators adjusted the video signs used in previous FIFA tournaments, which included the six internationally standardized video signs of potential sport-related concussions (in bold). Further signs were added and grouped into yellow and red flag categories.

If a yellow flag is observed, the injury spotter informs the FIFA Medical coordinator with details (including player team and number, mechanism of injury, and any video signs of possible concussion), and they will contact the team doctor with the recommendations for video review of the head impact and a clinical assessment. Further action will depend on the clinical assessment findings.

If a red flag is observed, the injury spotter informs the FIFA Medical coordinator with details, and they will strongly recommend immediate player substitution regardless of clinical assessment findings. The team doctor will be notified twice if the player is not substituted.

If no signs are observed, the FIFA medical coordinator is also notified. The team doctor is not notified unless they request further information.

The communication is recorded by the FIFA Medical Coordination/Injury spotter.

Yellow flags:

Lying motionless Lying without purposeful movement on the playing surface for >2 seconds. The player does not appear to move or react purposefully, respond or reply appropriately to the game situation (including team-mates, opponents, match officials or medical staff).

Blank/vacant look The player exhibits no facial expression or apparent emotion in response to the environment. This may include a lack of focus/attention of vision.

Disorientation The player appears to be disoriented in their movements and facial expressions.

Slow go get up The player takes longer than normal to rise to both feet after falling to the ground following a head impact.

Dual-head impact mechanism Two-immediate head impacts, such as head to ground impact after initial head-to-head impact.

Face or skull injury Any visible bleeding from the face or skull.

Red flags:

Impact seizure/convulsion Involuntary clonic movements that comprise periods of asymmetric and irregular rhythmic jerking of axial or limb muscles.

Tonic posturing Involuntary, sustained contraction of one or more limbs (typically upper limbs), so that the limb is held stiff despite the influence of gravity or the position of the player. Other muscles, such as the cervical, axial and lower-limb muscles, may also be involved. Tonic posturing may be observed while the player is on the playing surface or in the motion of falling, where the player may also demonstrate no protective action.

No protective action - Floppy The player falls to the playing surface in an unprotected manner (i.e. without stretching out their hands or arms to lessen or minimise the fall) after direct or indirect contact to the head. The player demonstrates loss of motor tone (which may be observed in the limbs and/or neck*) before landing on the playing surface.

*When the player's arms are being held by a tackling opponent, this may only be observed in the neck, which was previously known as "cervical hypotonia".

Motor incoordination The player appears unsteady on their feet (including losing balance, staggering/stumbling, struggling to get up or falling) or in the upper limbs (including fumbling). May occur when the athlete is rising from the playing surface or in the motion of walking/running.

Note: Should NOT be recorded if incoordination is considered related to an MSK injury (for example an ankle injury).

Vomiting Any immediate or delayed vomiting following head impact.

Visible concussive symptoms following return to play. Any symptoms of a brain injury following return to play after a head impact, such as confusion, impaired co-ordination, kneeling while clutching head or calling for team doctor re-assessment.

Other signs:

Concerning injury mechanism Obvious high head impact force, such as knee-to-head or fist-to-head. Location of head impact and head impact force (low/medium/high) should be recorded for all head impacts.

Uncontrolled emotional response Apparent exaggerated irritability/aggression either verbally or physically or crying.

Clutching of the head The player firmly presses or holds their head tightly immediately following head impact (rubbing the head with the hands is not considered clutching).

Additional video review After the tournament, broadcast video footage of all matches will be reviewed by an independent injury spotter, an athletic trainer with injury spotting training through Major League Soccer (MLS), and 1-2 years of experience with live injury spotting in MLS. The spotter will record all observed head impacts, mechanisms of injury, and identified observable signs, which will then be compared to those recorded during live action matches.

Video footage of each head impact, including the same video angles, which the injury spotter at the matches have access to, is then scored for video signs of concussion by three independent injury spotters blinded to each other's scoring.

Prior to review, these three injury spotters will perform inter-rater reliability testing of their identification of video signs in 20 head impacts from a set of exemplar signs selected from different competitions. A kappa value of minimum 0.8 will be required, and continuous discussion and rescoring will be performed until this is achieved.

For scoring of the included head impacts from the World Cup where there is not 100% agreement (3 of 3), there will be a review by an expert group to determine a final scoring.

Additionally, a sample of 10% of the incidents with full agreement will be reviewed by the expert group to ensure alignment on scoring.

The independent injury spotters will also record the head impact mechanism, location of the impact, presence and timing of medical assessment, whether there was foul play and sanction, and if the player was substituted, similar to a previous study.[9] Medical assessment is defined as any apparent clinical examination, direct talk, or visual inspection while the medical person is in close range of the player. Stoppage time is registered from when the ball is out of play, or the game is halted by the referee, following the head impact until the match is restarted.

Official match reports will be checked to determine whether a concussion substitution was used. The FIFA World Cup tournament follows protocol A of the IFAB additional permanent concussion substitution trial, where each team is allowed to use one concussion substitute in a match in addition to their normal substitutions.

The clinical diagnosis of a concussion will be recorded as part of the injury and illness surveillance at the FIFA World Cup, and included in this study if players have provided specific consent for this.

Statistics Simple descriptive statistics is applied using IBM SPSS Statistics for Windows (Version 27.0. Armonk, NY: IBM Corp) and results will be presented according to the distribution of the data.

Sample size estimation No a priori sample size calculation is performed. All head impacts will be included. Based on previous studies during football tournaments, we expect around 120-150 head impacts during the tournament, with up to half of these receiving on-pitch assessment by team medical staff.

ELIGIBILITY:
Inclusion Criteria:

* All participating football players at the FIFA World Cup Qatar 2022.

Exclusion Criteria:

* None

Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The FIFA World Cup Qatar 2022 includes 32 national teams, and each team is allowed to select 26 players, giving at total of 832 potential participants. In total, 64 matches will be played over 29 days.
Sampling Method: Non-Probability Sample
Enrollment: 832 (Actual)
Dates: Start 2022-11-20 (Actual); Primary Completion 2022-12-18 (Actual); Study Completion 2024-10-07 (Actual)

PRIMARY OUTCOMES:
Number of head impacts | November-December 2022
  A head impact is defined as '"a direct head impact, or impact with indirect forces to the head, where a player is unable to immediately resume play following impact or subsequently shows potential concussion-related symptoms."

SECONDARY OUTCOMES:
Number and type of video signs that indicate a potential concussion | November-December 2022
  Video signs are grouped as yellow or red flags. Yellow flags: Lying motionless Blank/vacant look Disorientation Slow go get up Dual-head impact mechanism Face or skull injury
  Red flags Impact seizure/ convulsion Tonic posturing No protective action Floppy
  Motor incoordination Vomiting Visible concussive symptoms following return to play.
  Other signs:
  Concerning injury mechanism Uncontrolled emotional response Clutching of the head
Head impact mechanism | November-December 2022
  Direct or indirect contact is categorised according to contact involved.
Location of the impact | November-December 2022
  The area of skull impact
presence and timing of medical assessments | November-December 2022
  Medical assessment is defined as any apparent clinical examination, direct talk, or visual inspection while the medical person is in close range of the player.
Foul play decisions | November-December 2022
  Referee decisions.
Presence of substitution following head impact | November-December 2022
  Official match reports will be check substitutions and to determine whether a concussion substitution was used.

CONTACTS AND LOCATIONS:
Locations (1):
- Major League Soccer, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared as it contains a high risk of exposing identifiable information.